CLINICAL TRIAL: NCT01178203
Title: The Effects of Three Oral Medications on Post-operative Pain Following Endodontic Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Peyman Mehrvarzfar, Department of Endodontics, Dental School of Tehran Azad University of Medical Sciences
Model: Parallel | Purpose: Treatment
Other Study IDs: IAU-1083
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-07

CONDITIONS: Pulpitis; Pain Management
Keywords: Endodontics; pain; visual analogue scale; NSAIDs
MeSH Terms: conditions — Pulpitis; Agnosia; Pain | interventions — Tramadol; L 5409709; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Placebo — Placebo
Drug: Tramadol — Tab, 100mg in 6, 12 and 24 hours after root canal treatment
Drug: Novafen — 325 mg in 6, 12 and 24 hours after root canal treatment
Drug: Naproxen — Tab, 500 mg in 6, 12, and 24 hours after root canal treatment

SUMMARY:
Aim: eliminating or reducing pain following endodontic treatment is of great importance. The aim of this study is to compare the effects of Tramadol, Novafen and Naproxen on post-operative pain following instrumentation of root canals in teeth with irreversible pulpitis. Sample size: one hundred patients considering the inclusion and exclusion criteria were selected. Intervention and outcome: The effect of Tramadol, Novafen and Naproxen on post-operative pain following instrumentation of root canals in teeth with irreversible pulpitis was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects were 20-60 years of age with no systemic diseases and females were not pregnant;
2. No history of taking any analgesics or other drugs prior to presenting for treatment;
3. Patients had moderate to severe pain associated with irreversible pulpitis in single-rooted premolars or anterior teeth.

Exclusion Criteria:

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 2010-07; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)